CLINICAL TRIAL: NCT06356051
Title: Evaluation of Cardiovascular Disease Risk in Children With Type 1 Diabetes Mellitus by Oscillometric Method and Echocardiography
Brief Title: Cardiovascular Disease Risk in Children With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: Gbuyukyilmaz
Record Dates: First submitted 2024-03-25; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type1 diabetes mellitus
  Interventions: Device: Echocardiography
- Healthy children
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — cardiovascular evaluation
  Other Names: oscillometric Mobil-O-Graph device

SUMMARY:
Epicardial fat thickness, carotid intima-media thickness, and augmentation index from arterial stiffness indicators are increased in children with T1DM compared to the healthy control group. These results support the idea that children with T1DM present significant changes in important subclinical indicators for the development of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. type T1DM patients
2. body mass index (BMI) between the 5th and 85th percentile according to age and gender
3. having T1DM for at least 2 years
4. ages 8-18 years

Exclusion Criteria:

1. having any chronic diseases other than T1DM
2. presence of a congenital and/or acquired heart disease, hypertension etc.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: type 1 diabetes mellitus and age and gender mathced healthy children
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Epicardial fat thickness | january 2023-june 2023
  Epicardial fat thickness was measured with Echocardiography as milimeter. Epicardial fat was identified as the echo-free space between the outer wall of the myocardium and the visceral layer of pericardium. The values of children with type 1 DM were compared with healthy children. Values are given as mean and standard deviation.

SECONDARY OUTCOMES:
carotid intima-media thickness | january 2023-june 2023
  carotid intima-media thickness were measured by echocardiography machine as milimeter. cIMT is defined as the distance between the first echogenic line (lumen-intima interface) and the second echogenic line (media-adventitia interface) of the far wall. The values of children with type 1 DM were compared with healthy children. Values are given as mean and standard deviation.
arterial stiffness parameters such as pulse wave velocity, augmentation index | january 2023-june 2023
  cuff-based validated oscillometric Mobil-O-Graph device (I.E.M., GmbH, Aachen, Germany) was used to these parameters. Data from the Mobil-O Graph device was exported and analyzed using Hypertension Management Software Client-Server version 5.2.3. The values of children with type 1 DM were compared with healthy children. Values are given as mean and standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT06356051/Prot_SAP_000.pdf